CLINICAL TRIAL: NCT05846399
Title: CAT BITE Antibiotic Prophylaxis and Durations for the Hand/Forearm (CATBITE): A Prospective, Randomized, Placebo-controlled, Double-blinded, Clinical Trial
Brief Title: CAT BITE Antibiotic Prophylaxis for the Hand/Forearm (CATBITE)
Acronym: CATBITE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Stephen Colbert, CHIEF OF DIVISION OF PLASTIC SURGERY AND PROFESSOR OF SURGERY, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2092043
Record Dates: First submitted 2023-04-12; First posted 2023-05-06 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Cat Bite; Hand Injuries; Arm Injury; Infection, Bacterial; Anti-bacterial Agents
MeSH Terms: conditions — Hand Injuries; Arm Injuries; Bacterial Infections | interventions — Amoxicillin-Potassium Clavulanate Combination; Ciprofloxacin; Clindamycin; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Placebo-controlled, Double-blinded, Clinical Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: A double-blinded protocol will be performed. Investigators and participants will be blinded to study interventions. Both will be blinded to reduce the risk of bias. All three interventions will be packaged in identical capsule vials. The placebo arm will have all capsules filled with microcrystalline cellulose and no active drug, the one day intervention arm will be packaged in identical capsule vials with the first day of active drug and four days filled with placebo, five day intervention group will be packaged in identical capsule vials with all capsules filled with active drug. Blinding will remain throughout the duration of the study. Following completion of patient participation (day 30+/-2). Investigators and participants will be notified of the respective treatment arms. Final results will be available to investigators and participants following completion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (microcrystalline cellulose) (Placebo Comparator): Placebo capsules by mouth twice daily x 5 days (5 days of placebo microcrystalline cellulose capsules)
  Interventions: Other: Placebo (microcrystalline cellulose); Procedure: Wound management
- Antibiotic x 1 day (Active Comparator): Amoxicillin-clavulanate 875-125mg capsules by mouth twice daily x 1 day (4 days of placebo capsules)
  -Penicillin allergy: ciprofloxacin 500mg by mouth twice daily + clindamycin 300mg by mouth three times daily x 1 day
  Interventions: Drug: Amoxicillin/clavulanate; Drug: Ciprofloxacin; Drug: Clindamycin; Other: Placebo (microcrystalline cellulose); Procedure: Wound management
- Antibiotic x 5 days (Active Comparator): Amoxicillin-clavulanate 875-125mg capsules by mouth twice daily x 5 days (0 days of placebo capsules)
  -Penicillin allergy: ciprofloxacin 500mg by mouth twice daily + clindamycin 300mg by mouth three times daily x 5 days
  Interventions: Drug: Amoxicillin/clavulanate; Drug: Ciprofloxacin; Drug: Clindamycin; Procedure: Wound management

INTERVENTIONS:
Drug: Amoxicillin/clavulanate — Amoxicillin-clavulanate 875-125mg by mouth twice daily for 1 day or Ciprofloxacin 500mg by mouth twice daily and clindamycin 450mg by mouth twice daily for 1 day
  Other Names: Augmentin; Clavulin; Betacillin; Clavamox
  Arms: Antibiotic x 1 day; Antibiotic x 5 days
Drug: Ciprofloxacin — Amoxicillin-clavulanate 875-125mg by mouth twice daily for 5 days or Ciprofloxacin 500mg by mouth twice daily and clindamycin 450mg by mouth twice daily for 5 days
  Other Names: Cipro
  Arms: Antibiotic x 1 day; Antibiotic x 5 days
Drug: Clindamycin — Amoxicillin-clavulanate 875-125mg by mouth twice daily for 5 days or Ciprofloxacin 500mg by mouth twice daily and clindamycin 450mg by mouth twice daily for 5 days
  Other Names: Cleocin
  Arms: Antibiotic x 1 day; Antibiotic x 5 days
Other: Placebo (microcrystalline cellulose) — Placebo (microcrystalline cellulose) by mouth twice daily by mouth for 5 days
  Other Names: (C6H10O5)n
  Arms: Antibiotic x 1 day; Placebo (microcrystalline cellulose)
Procedure: Wound management — Wound management includes hemostasis, copious irrigation, removal of foreign bodies, and excisional debridement of devitalized tissue. If only punctures are present, lancing of the punctures is not typically required unless infection has already developed. Local anesthesia (1% lidocaine hydrogen chloride (HCl) with epinephrine 1:100,000; 200mg/20mL vial) will be used prior to irrigation (30mL of povidone-iodine in 1L of 0.9% sodium chloride (NaCl) solution and/or 118mL of 3% hydrogen peroxide) and debridement. Open wounds will be irrigated and debrided at bedside. Wounds will be covered with soft dressings in place until first follow-up at day 2.

SUMMARY:
Cat bites are puncture wounds that have the potential to seed bacteria deep within the joint capsule, periosteum, and bone. The hand is the most common site of bite injuries. Pasteurella multocida is the is the most common organism isolated from the mouths of cats that can cause infections after a bite. Prophylactic antibiotics are often recommended with amoxicillin-clavulanate for 3-5 days to decrease the incidence of developing an infection. However, only one randomized controlled clinical trial consisting of 12 patients has been performed to justify this course of treatment, raising the possibility that the use of antibiotics could be reduced or even eliminated. Investigators will compare different durations of prophylactic antibiotics and a placebo control for cat bites to the hand/forearm presenting to the Emergency Department, Urgent Care, Plastic Surgery Clinic using a randomized, controlled, double-blind clinical trial. Participants presenting to the University of Missouri Hospital Emergency Department, Missouri University (MU) Healthcare Urgent Care, Plastic Surgery Clinic over the next year will be offered the chance to enroll if they meet the inclusion/exclusion criteria. For inclusion, participants will be >18 years of age, have cat bites to the hand or distal to elbow, and present within 24 hours of the cat bite injury. Participants must not present with active local or systemic infections, have received antibiotics within the past 30 days, or be immunocompromised (primary and secondary immunodeficiencies). Participants will be randomized to one of three treatment arms (placebo; amoxicillin-clavulanate 1 day; amoxicillin-clavulanate 5 days). Outcomes are the development of an infection at the location of the cat bite and/or systemic infection, adverse effects of interventions, disability assessed by Quick Disabilities of Arm, Shoulder and Hand (QuickDASH) scores, and quality of life (QOL) assessed by HAND Questionnaire (HAND-Q) scores. Infection will be assessed at day 0, day 2, day 7+/-2, day 14+/-2, and day 30+/-2 by vital signs, laboratory values, physical examination and with an infrared and digital camera. All measures will be within the standard of care, apart from the infrared camera, QuickDASH, and HAND-Q scores. The anatomic locations of cat bites to the hand/forearm will be assessed for correlations with infections.

DETAILED DESCRIPTION:
Cat bites have been reported as the second most common domestic animal bite in the United States, ranging from 5%-15% of all bites. The hand is the most common site of bite injuries. Cat bites are puncture wounds that have the potential to seed bacteria deep within the joint capsule, periosteum and bone. As a result, infection is a serious complication, reported in 30%-50% of cat bites. The median time to signs and symptoms of infection following a cat bite is typically short (approximately 12 hours). Direct healthcare costs associated with management of cat and dog bites in the United States estimate >$850,000,000 annually and do not consider the indirect costs associated with time off work, rehabilitation, and permanent impairment.

The average cat bite wound culture yields five types of bacterial isolates. Mixed aerobic and anaerobic bacteria are observed in 60% of cases. Pasteurella multocida is the is the most common organism isolated from the mouths of cats that can cause infections after a bite. Pasteurella species are isolated from 75% of cat bite wounds, and the incubation period for Pasteurella infection is one to three days. Capnocytophaga canimorsus can cause bacteremia and fatal sepsis after animal bites, especially in patients with asplenia, alcoholism, or underlying hepatic disease. The incubation period for Capnocytophaga infection is one to three days. Bartonella henselae may be transmitted via the bite of an infected cat and contact with cat saliva via broken skin or mucosal surfaces. The incubation period for Bartonella infection is 7 to 14 days. Anaerobes isolated from dog and cat bite wounds include Bacteroides species, fusobacteria, Porphyromonas species, Prevotella species, cutibacteria (formerly propionibacteria), and peptostreptococci.

Prophylactic antibiotics are often recommended to decrease the incidence of developing an infection. Broad antibiotic coverage is recommended to address the polymicrobial nature of common oral flora and bite infections. Pasteurella species are generally susceptible to penicillin and ampicillin, but staphylococci and anaerobic species often produce beta-lactamase, which provides resistance to these antibiotics. Adding a beta-lactamase inhibitor significantly increases the effectiveness of these antibiotics, and amoxicillin-clavulanate is the oral antibiotic of choice for human, dog, and cat bites. Infectious Diseases Society of America (IDSA) guidelines recommend antibiotic prophylaxis with amoxicillin-clavulanate 875-125mg twice daily (BID) for 3-5 days or ciprofloxacin 500-750mg BID + clindamycin 300-450mg three times daily (TID) if a participant has a penicillin allergy. However, only one randomized controlled clinical trial (RCT) has been performed to date to assess the efficacy of prophylactic antibiotics following cat bites. Adult participants with uninfected full-thickness wounds presenting within 24 hours of injury to the emergency department were considered. Participants were randomly assigned to receive oxacillin 500mg four times daily (QID) for five days (n=5) or identically appearing placebo (n=6). Four of six participants receiving placebo, but none of the five participants receiving oxacillin, developed a wound infection (P = 0.045).

Immunocompetent adult participants presenting within 24 hours of a cat bite without any signs or symptoms of infection may benefit from advances in wound care alone or only need a maximum of 24 hours of antibiotic prophylaxis. Furthermore, a Cochrane review aggregating data from clinical trials from the literature concluded, "There is no evidence that the use of prophylactic antibiotics is effective for cat or dog bites." The investigators' hypothesis is that administration of 5 days of prophylactic antibiotics will not reduce the incidence of infection in participants evaluated and treated within 24 hours of cat bite injury, who do not exhibit signs of an active infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater or equal to 18 years of age.
* Bitten by a cat.
* Location of bite is the hand and/or forearm (distal to elbow).
* Presenting <24 hours following a cat bite to the hand/forearm.
* English speaking

Exclusion Criteria:

* Patients who present with active local or systemic infections

  1. Purulent drainage from the cat bite
  2. Redness AND swelling at the location of the cat bite
* Having a fever >100.4° F or >38° C)-Received antibiotics within the past 30 days
* Received antibiotics within the past 30 days
* Patients unwilling to take study medication
* Patients unwilling to attend scheduled follow-up evaluations or complete study forms
* Pregnant Women
* Type I hypersensitivity reaction to any of the study interventions
* Immunocompromised patients (primary and secondary immunodeficiencies) Primary
* Autoimmune Lymphoproliferative Syndrome (ALPS)
* Autoimmune Polyglandular Syndrome type 1 (APS-1)
* B-cell Expansion with Nuclear factor kappa-light-chain-enhancer of activated B cells and T-cell Anergy (BENTA) Disease
* Caspase Eight Deficiency State (CEDS)
* Caspase Recruitment Domain Family Member 9 (CARD9) Deficiency and Other Syndromes of Susceptibility to Candidiasis
* Cartilage-hair hypoplasia
* Chédiak-Higashi syndrome
* Chronic Granulomatous Disease (CGD)
* Common Variable Immunodeficiency (CVID)
* Complement Deficiencies
* Congenital Neutropenia Syndromes
* Cytotoxic T-Lymphocyte Associated Protein 4 (CTLA4) Deficiency
* Cyclic neutropenia
* DiGeorge syndrome
* Dedicator Of Cytokinesis 8 (DOCK8) Deficiency
* GATA-binding protein 2 (GATA2) Deficiency
* Glycosylation Disorders with Immunodeficiency
* Hyper-Immunoglobulin E Syndromes (HIES)
* Hyper-Immunoglobulin M Syndromes
* Interferon Gamma, Interleukin 12 and Interleukin 23 Deficiencies
* Leukocyte Adhesion Deficiency (LAD) Types 1 and 2
* Lipopolysaccharide Responsive Beige-Like Anchor Protein (LRBA) Deficiency
* Phosphatidylinositol 3-kinase (PI3-Kinase) Disease
* Phospholipase C gamma 2 (PLCG2) associated Antibody Deficiency and Immune Dysregulation (PLAID)
* Severe Combined Immunodeficiency (SCID)
* Selective Immunoglobulin A (IgA) deficiency
* Signal transducer and activator of transcription 3 (STAT3) Dominant-Negative Disease
* STAT3 Gain-of-Function Disease
* Warts, Hypogammaglobulinemia, Infections, and Myelokathexis (WHIM) Syndrome
* Wiskott-Aldrich Syndrome (WAS)
* X-Linked Agammaglobulinemia (XLA)
* X-Linked Lymphoproliferative Disease (XLP)
* X-linked magnesium transporter 1 (MAGT1) deficiency with increased susceptibility to Epstein-Barr virus (EBV) infection and N-linked glycosylation defect (XMEN) Disease
* Zeta-associated protein 70 (ZAP-70) deficiency

Secondary

* Malnutrition
* Uncontrolled Diabetes mellitus
* Chronic uremia
* Genetic syndromes: trisomy 21
* Immunomodulatory, immunosuppressive drug therapy: corticosteroids, calcineurin inhibitors, cytotoxic agents
* Systemic lupus erythematosus
* Malignancy
* Active radiation therapy
* Bone marrow ablation
* Infectious diseases: human immunodeficiency virus (HIV) infection, Hepatitis

Additional Primary and secondary immunodeficiencies can be found at the following link.

https://www.merckmanuals.com/professional/immunology-allergic-disorders/immunodeficiency-disorders/overview-of-immunodeficiency-disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of infection | Day 30+/-2
  To compare the incidence of infection (skin, soft tissue, joint, bone) between each study arm to determine the effect of antibiotic prophylaxis and duration on cat bites to the hand and/or forearm within 30 days. Infections are defined by, The Centers for Disease Control and Prevention National Healthcare Safety Network.
Changes of the incidence of infection | Day 2; Day 7+/-2; Day 14+/-2; Day 30+/-2
  To compare changes of the incidence of infection (skin, soft tissue, joint, bone) between each study arm and within each study arm to determine the effect of antibiotic prophylaxis and duration on cat bites to the hand and/or forearm at different time points. Infections are defined by the The Centers for Disease Control and Prevention National Healthcare Safety Network.

SECONDARY OUTCOMES:
Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) scores | Day 30+/-2
  To compare QuickDASH scores between each study arm to determine the effect of antibiotic prophylaxis and duration on a patient's disability following cat bites to the hand and/or forearm within 30 days. different time points. QuickDASH scores are measured on a scale of 0 to 100 (higher scores indicate increased patient-reported disability).
Changes in Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) scores | Day 0, Day 2; Day 7+/-2; Day 14+/-2; Day 30+/-2
  To compare changes in QuickDASH scores between each study arm and within each study arm to determine the effect of antibiotic prophylaxis and duration on a patient's disability following cat bites to the hand and/or forearm at different time points. QuickDASH scores are measured on a scale of 0 to 100 (higher scores indicate increased patient-reported disability).
HAND Questionnaire (HAND-Q) scores | Day 30+/-2
  To compare HAND-Q scores between each study arm to determine the effect of antibiotic prophylaxis and duration on a patient's quality of life following cat bites to the hand and/or forearm within 30 days. The HAND-Q is composed of independently functioning scales scored separately. To score a scale, the raw scores for the set of items in a scale are added together to produce a total raw score. Items are summed to produce a total scale raw score. A conversion table is used to convert raw scores into a score that ranges from 0 (worst) to 100 (best). The conversion, which linearizes the scores, is based on the findings from the Rasch analysis. Higher scores for HAND-Q scales reflect a better outcome.
Changes in HAND Questionnaire (HAND-Q) scores | Day 0, Day 2; Day 7+/-2; Day 14+/-2; Day 30+/-2
  To compare changes in HAND-Q scores between each study arm and within each study arm to determine the effect of antibiotic prophylaxis and duration on a patient's quality of life following cat bites to the hand and/or forearm at different time points. The HAND-Q is composed of independently functioning scales scored separately. To score a scale, the raw scores for the set of items in a scale are added together to produce a total raw score. Items are summed to produce a total scale raw score. A conversion table is used to convert raw scores into a score that ranges from 0 (worst) to 100 (best). The conversion, which linearizes the scores, is based on the findings from the Rasch analysis. Higher scores for HAND-Q scales reflect a better outcome.
Adverse effects | Day 30+/-2
  To compare adverse effects between each study arm to determine the adverse effects of antibiotic prophylaxis and duration on cat bites to the hand and/or forearm within 30 days.
Changes in adverse effects | Day 0, Day 2; Day 7+/-2; Day 14+/-2; Day 30+/-2
  To compare changes in adverse effects between each study arm and within each study arm to determine the adverse effects of antibiotic prophylaxis and duration on cat bites to the hand and/or forearm at different time points.

OTHER OUTCOMES:
Location of cat bites that result in infection | Day 30+/-2
  To determine if the anatomic location of the cat bite results in the development of the infection within 30 days.
Changes in location of cat bites that result in infection | Day 0, Day 2; Day 7+/-2; Day 14+/-2; Day 30+/-2
  To determine if the anatomic location of the cat bite between each study arm and within each study arm results in the development of the infection at different time points.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Klifto, DO, PharmD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with researchers who have not been approved as study members by the University of Missouri IRB

REFERENCES:
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Background] Sierakowski K, Dean NR, Pusic AL, Cano SJ, Griffin PA, Bain GI, Klassen A, Lalonde D. International multiphase mixed methods study protocol to develop a cross-cultural patient-reported outcome and experience measure for hand conditions (HAND-Q). BMJ Open. 2019 Mar 20;9(3):e025822. doi: 10.1136/bmjopen-2018-025822. PMID 30898824
- [Background] Bregman B, Slavinski S. Using emergency department data to conduct dog and animal bite surveillance in New York City, 2003-2006. Public Health Rep. 2012 Mar-Apr;127(2):195-201. doi: 10.1177/003335491212700208. PMID 22379219
- [Background] Kwo S, Agarwal JP, Meletiou S. Current treatment of cat bites to the hand and wrist. J Hand Surg Am. 2011 Jan;36(1):152-3. doi: 10.1016/j.jhsa.2009.10.008. Epub 2009 Dec 14. No abstract available. PMID 20006917
- [Background] Benson LS, Edwards SL, Schiff AP, Williams CS, Visotsky JL. Dog and cat bites to the hand: treatment and cost assessment. J Hand Surg Am. 2006 Mar;31(3):468-73. doi: 10.1016/j.jhsa.2005.12.011. PMID 16516744
- [Background] Kennedy SA, Stoll LE, Lauder AS. Human and other mammalian bite injuries of the hand: evaluation and management. J Am Acad Orthop Surg. 2015 Jan;23(1):47-57. doi: 10.5435/JAAOS-23-01-47. PMID 25538130
- [Background] Talan DA, Citron DM, Abrahamian FM, Moran GJ, Goldstein EJ. Bacteriologic analysis of infected dog and cat bites. Emergency Medicine Animal Bite Infection Study Group. N Engl J Med. 1999 Jan 14;340(2):85-92. doi: 10.1056/NEJM199901143400202. PMID 9887159
- [Background] Medeiros I, Saconato H. Antibiotic prophylaxis for mammalian bites. Cochrane Database Syst Rev. 2001;(2):CD001738. doi: 10.1002/14651858.CD001738. PMID 11406003
- [Background] Lloret A, Egberink H, Addie D, Belak S, Boucraut-Baralon C, Frymus T, Gruffydd-Jones T, Hartmann K, Hosie MJ, Lutz H, Marsilio F, Mostl K, Pennisi MG, Radford AD, Thiry E, Truyen U, Horzinek MC. Pasteurella multocida infection in cats: ABCD guidelines on prevention and management. J Feline Med Surg. 2013 Jul;15(7):570-2. doi: 10.1177/1098612X13489215. PMID 23813817
- [Background] Stevens DL, Bisno AL, Chambers HF, Everett ED, Dellinger P, Goldstein EJ, Gorbach SL, Hirschmann JV, Kaplan EL, Montoya JG, Wade JC; Infectious Diseases Society of America. Practice guidelines for the diagnosis and management of skin and soft-tissue infections. Clin Infect Dis. 2005 Nov 15;41(10):1373-406. doi: 10.1086/497143. Epub 2005 Oct 14. No abstract available. PMID 16231249
- [Background] Coburn B, Toye B, Rawte P, Jamieson FB, Farrell DJ, Patel SN. Antimicrobial susceptibilities of clinical isolates of HACEK organisms. Antimicrob Agents Chemother. 2013 Apr;57(4):1989-91. doi: 10.1128/AAC.00111-13. Epub 2013 Feb 12. PMID 23403420
- [Background] Beasley H, Borgmann AR, McDonald TO, Belluscio PR. Carbachol in cataract surgery. Arch Ophthalmol. 1968 Jul;80(1):39-41. doi: 10.1001/archopht.1968.00980050041006. No abstract available. PMID 5660015
- [Background] Elenbaas RM, McNabney WK, Robinson WA. Evaluation of prophylactic oxacillin in cat bite wounds. Ann Emerg Med. 1984 Mar;13(3):155-7. doi: 10.1016/s0196-0644(84)80604-6. PMID 6696302